CLINICAL TRIAL: NCT06658470
Title: Investigation of the Turkish Validity and Reliability of Hand Disability In Systemic Sclerosis - Digital Ulcersthe (HDISS-DU) Questionnaire in Individuals With Systemic Sclerosis
Brief Title: Hand Disability In Systemic Sclerosis - Digital Ulcers
Status: Enrolling by invitation | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Zülal TATAR, Researcher, Pamukkale University
Other Study IDs: SSc Validity and Reliability
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-10

CONDITIONS: Systemic Sclerosis (SSc); Digital Ulcer
MeSH Terms: conditions — Scleroderma, Systemic; digital ulcers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study was to examine the Turkish validity and reliability of the Hand Disability in Systemic Sclerosis - Digital Ulcers Questionnaire (HDISS-DU) in individuals with Systemic Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SSc by a rheumatologist
* Being 18 years of age or older

Exclusion Criteria:

* Presence of neurological disease
* Presence of any orthopedic problem that would affect functionality
* Presence of a history of orthopedic surgery
* Inability to speak or understand Turkish fluently
* Presence of a psychiatric disease that would affect cooperation
* Severe neurological disease that would affect hand functions (peripheral nerve lesion, trauma, operation, cerebrovascular accident)
* Heart failure and lung pathology that would affect daily living activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include individuals aged 18 and older who are receiving treatment for Systemic Sclerosis at two university hospital in Turkey, and meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
The Hand Disability in Systemic Sclerosis-Digital Ulcers Questionnaire | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  It was developed to evaluate the disability caused by digital ulcers in the hand in patients with Systemic Sclerosis. It consists of 24 questions. There are 8 response options. Responses are scored from 1 to 6. 1 'yes, without difficulty'; 2 'yes, with very little difficulty', 3 'yes, with some difficulty', 4 'yes, with great difficulty', 5 'almost impossible' and 'using only the unaffected hand' (same score for both responses) and 6 'impossible'. The eighth response option 'did not do this activity in the last 7 days' is not included in the scoring. The total HDISS-DU score is calculated as the average of the scores of the questions where the eighth option was not given as an answer (threshold for questions with an eighth answer <12 questions). The total score ranges from a minimum of 1 point to a maximum of 6 points.

SECONDARY OUTCOMES:
Scleroderma Health Assessment Questionnaire | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Used to assess disease activity. It has 20 items in 8 sections assessing physical disability. In addition, Raynaud phenomenon, digital ulcers, pulmonary and gastrointestinal symptoms are assessed according to the Visual Analog Scale, which is scored between "0" and "10". VAS is scored between 0 and 3 by multiplying by 0.2
Cochin 17-Item Scleroderma Functional Scale | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  The scle assesses activity and participation in patients with systemic sclerosis. It consists of 17 items and two sections: Section A (10 items, factor 1) assesses mobility. Section B (7 items, factor 2) assesses general tasks and demands. The score for each section is the sum of the scores for each item: Section A scores range from 0 to 100, and Section B scores range from 0 to 70. The total score for the Cochin 17-Item Scleroderma Functional Scale is defined as the sum of the scores for each section and ranges from 0 (no limitation) to 170 (maximum limitation).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Pamukkale University, Denizli, Malatya
  - Inonu University, Malatya, Malatya